CLINICAL TRIAL: NCT04117737
Title: Effects of Virtual Reality Combined With Antigravity Treadmill Rehabilitation for Gait Improvement of Patients With Parkinson's Disease: a Pilot Study
Brief Title: A Pilot Study of Virtual Reality and Antigravity Treadmill for Gait Improvement in Parkinson
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI18/386
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2019-12

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic
Keywords: Parkinson; Virtual reality; Anti-gravity treadmill; Rehabilitation; Gait disorders
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic; Mobility Limitation

STUDY DESIGN:
Masking Description: Outcomes assessor was blinded to outcomes values between sessions and to the adherence of participants to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Single-arm
  Interventions: Other: Virtual reality combined with anti-gravity treadmill

INTERVENTIONS:
Other: Virtual reality combined with anti-gravity treadmill — The system is composed of three major parts: the treadmill, the antigravity system and the virtual reality system.
  The treadmill is the base of the device. It is a rounded and concave structure that permits to walk in all direction. For simulate anti-gravity, a harness and pulley system allow to regulate the weight. Finally, the virtual reality system enables participants to simulate an experience of daily life.

SUMMARY:
The aim of this study is to improve knowledge about mechanical gait assistance combined with virtual reality efficiency in gait recovery for Parkinson´s patients. It is hypothesised that 12 sessions of 30 minutes each, over a 4 weeks period, of antigravity treadmill rehabilitation combined with virtual reality treatment is effective for increase gait autonomy in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Having Parkinson's disease diagnosed by a neurological doctor.
* Having an alteration of the gait caused by the neurological disorder.
* Being able to have an independent and voluntary walk of 10 meters as minimum.
* Height more than 150 cm.

Exclusion Criteria:

* Being blind.
* Medical contraindications for walking.
* Being amputee.
* Alcohol or drugs abuse.
* Other diseases that impedes the intervention.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in gait autonomy | Baseline and 4-weeks
  Changes in gait autonomy will be measured by 6-Minutes Walking Test (6MWT). The 6MWT consists of measuring the maximum distance (in meters) that the subject can walk during 6 minutes in a flat surface.

SECONDARY OUTCOMES:
Changes in gait speed | Baseline and 4-weeks
  Changes in gait speed will be measured by 10-Meter Walk Test (10MWT). The 10MWT consists of asking the subject to walk a 14m distance on flat area and measure the time spent from meter 2 to meter 12. Time will be measured by a digital chronometer. Gait speed will be calculated in meter per second.
Changes in balance and gait ability | Baseline and 4-weeks
  Changes in balance and gait ability will be measured by Tinetti scale. The Tinetti test is a simple, reproducible way of assessing the risk of falling in the elderly. This scale is composed of two value, static and dynamic: the test grants a maximum of 16 points for static part (sitting) and 12 point for dynamic (walking) part. Higher is the score, better is the performance.
Changes in quality of life | Baseline and 4-weeks
  Changes in quality of life will be measured by by 36-Item Short-Form Health Survey (SF-36). SF-36 assesses 8 physical and mental health domains: 1) Physical Functioning, 2) Social Functioning, 3) Role-Physical, 4) Bodily Pain, 5) Mental Health), 6) Role-Emotional, 7) Vitality, and 8) General Health. For each scale, item scores are coded, summed, and transformed, with final values expressed as a percentage, ranging from 0 (worst health) to 100 (best health).

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Herrero, PhD, Principal Investigator — Universidad San Jorge
Locations (1):
- Asociación de Parkinson de Aragón, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No
There are currently no plan on sharing data from this study with other researchers.